CLINICAL TRIAL: NCT02761187
Title: A Global, Prospective, Non-interventional, Observational Study of Presentation, Treatment Patterns, and Outcomes in Multiple Myeloma Patients - the INSIGHT - MM Study
Brief Title: An Observational Study of Presentation, Treatment Patterns, and Outcomes in Multiple Myeloma Participants
Status: Terminated | Type: Observational
Why Stopped: This study was stopped 3 years early due to business reprioritization within Takeda
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: NSMM-5001
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newly Diagnosed Multiple Myeloma: Participants newly diagnosed with MM within 3 months from initiation of treatment were enrolled for 3 years, and followed for at least 2 years, until death, or the end of the study, whichever comes first (up to approximately 5 years).
  Interventions: Other: No Intervention
- Relapsed/Refractory Multiple Myeloma: Participants diagnosed with RRMM who previously received 1 to 3 prior lines of therapy were enrolled for 3 years, and followed for at least 2 years, until death, or the end of the study, whichever comes first (up to approximately 5 years).
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this was an observational study, no intervention was administered.

SUMMARY:
The purpose of this study is to describe contemporary, real-world patterns of participant characteristics, clinical disease presentation, therapeutic regimen chosen, and clinical outcomes in participants with newly diagnosed [ND] multiple myeloma (MM) and participants with relapsed/refractory [R/R] MM.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, observational study. This study will look at contemporary, real-world patterns of participant characteristics, clinical disease presentation, therapeutic regimen chosen, and clinical outcomes in participants with MM. Participants will not be asked to change their routine clinical treatment. Participants will have to complete patient reported outcomes (PROs) surveys during on-site routine office visits.

The study will enroll approximately 4200 participants. Participants will be assigned to one of the following cohorts based upon the diagnosis of MM:

* ND MM within 3 months from initiation of treatment
* R/R MM who have received 1 to 3 prior lines of therapy

This multi-center trial will be conducted worldwide. The overall time to participate in this study is up to 8 years. Participants will be evaluated and followed-up for a period of at least 5 years, until death, are lost to follow-up, or the end of the study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

Is 18 years of age or older.

Is experiencing the following:

1. Newly diagnosed MM within 3 months from initiation of treatment with documented month and year of diagnosis, criteria met for diagnosis, stage, and MM-directed treatment history, including duration, or
2. Relapsed/refractory MM who have received 1 to 3 prior lines of therapy with documented data in the medical record regarding diagnosis (month and year), the regimens used in 1st, 2nd, and 3rd line as applicable, whether stem cell transplant was part of 1st, 2nd, and 3rd line of therapy, whether consolidation/maintenance was part of 1st, 2nd, and 3rd line of therapy, also whether investigational therapy/treated on a clinical trial was part of any of these regimens.

Is willing and able to sign informed consent to participate. Is willing and able to complete patient-reported outcomes (PROs) in accordance with local regulatory and data protection requirements.

Exclusion Criteria:

Is reporting to a site in this study for a second opinion (consultation only) or participants whose frequency of consult and follow-up are not adequate for quarterly electronic case report form (eCRF) completion.

Has participated in another study (observational or interventional) that prohibits participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Multiple Myeloma
Sampling Method: Probability Sample
Enrollment: 4253 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (137):
- United States (43):
  - CARTI Cancer Center, Little Rock, Arkansas
  - University of Arkansas For Medical Sciences, Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Rocky Mountain Cancer Centers (Williams) - USOR, Denver, Colorado
  - Poudre Valley Health System, Fort Collins, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - SCRI Florida Cancer Specialists East, Daytona Beach, Florida
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - SCRI Florida Cancer Specialists North, St. Petersburg, Florida
  - Illinois Cancer Specialists (Niles) - USOR, Niles, Illinois
  - Indiana University, Indianapolis, Indiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Maryland Oncology Hematology (Columbia) - USOR, Columbia, Maryland
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Central Care Cancer Center, Bolivar, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Saint Francis Hospital, East Hills, New York
  - Mount Sinai Medical Center, New York, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Hematology Oncology Associates - USOR, Medford, Oregon
  - Northwest Cancer Specialists (Broadway) - USOR, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - SCRI Tennessee Oncology Nashville, Nashville, Tennessee
  - Texas Oncology (Loop) - USOR, Amarillo, Texas
  - Texas Oncology (Loop) - USOR, Dallas, Texas
  - Texas Oncology (Loop) - USOR, El Paso, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology (Loop) - USOR, Round Rock, Texas
  - Texas Oncology (Loop) - USOR, San Antonio, Texas
  - Yakima Valley Memorial Hospital North Star Lodge - USOR, Yakima, Washington
  - Berkeley Medical Center, Martinsburg, West Virginia
  - St Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Milwaukee, Wisconsin
- Belgium (6):
  - Grand Hopital de Charleroi asbl, Charleroi
  - UZ Gent, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - UZ Leuven, Leuven
  - CHU de Liege, Liège
  - CHU UCL Namur asbl - Site Godinne, Yvoir
- Brazil (8):
  - Unicamp Universidade Estadual de Campinas, Campinas
  - Centro de Pesquisas Oncologicas, Florianópolis
  - Hospital Das Clinicas Da Universidade Federal de Goias, Goiânia
  - Universidade Federal Do Rio de Janeiro Hospital Universitario Clementino Fraga Filho, Rio de Janeiro
  - CEHON - Centro de Hematologia e Oncologia da Bahia Ltda, Salvador
  - Clinica Sao Germano, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- China (4):
  - Peking Union Medical College Hospital, Beijing
  - Peking University Peoples Hospital, Beijing
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - First Affiliated Hospital of Soochow University, Suzhou
- Colombia (4):
  - Fundacion Santa Fe de Bogota, Bogotá
  - Fundacion Oftalmologica de Santander Foscal, Floridablanca
  - Hospital Pablo Tobon Uribe, Medellín
  - Oncomedica SA, Montería
- France (6):
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier de Perigueux, Périgueux
  - CHRU de Poitiers La Miletrie, Poitiers
  - CHU de Nancy-Hopital Brabois Adulte, Vandœuvre-lès-Nancy
- Germany (10):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Gefos - Gesellschaft fur onkologische Studien mbH, Dortmund
  - Universitatsklinikum Heidelberg, Heidelberg
  - Internistisch Hamatologische und Internistische Praxis, Herrsching am Ammersee
  - Institut fur Versorgungsforschung in der Onkologie GbR, Koblenz
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz
  - Mannheimer Onkologie Praxis, Mannheim
  - OnkoNet Marburg GmbH, Marburg
  - Onkologische Gemeinschaftspraxis Siegburg, Siegburg
  - Universitatsklinikum Tubingen, Tübingen
- Greece (6):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Evangelismos General Hospital of Athens, Athens
  - Alexandra Hospital, Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - University General Hospital of Patras, Pátrai
- Israel (6):
  - HaEmek Medical Center, Afula
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kefar Sava
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Medical Centers, Tel Aviv
- Italy (8):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G.M. Lancisi G. Salesi, Ancona
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Policlinico Umberto I, Roma
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
- Mexico (4):
  - Nucleo Oncologico de Occidente S.C., Guadalajara
  - Hematologica Alta Especialidad S.C., Huixquilucan
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey
- Spain (6):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Complejo Asistencial Universitario de Leon, León
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Taiwan (6):
  - Chang Gung Medical Foundation Chiayi Chang Gung Memorial Hospital, Buzi, Chiayi County
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (10):
  - Cukurova Universitesi Tip Fakultesi Balcali Hastanesi, Adana
  - Ankara University Medical Faculty Cebeci Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Johns Hopkins Medicine - Anadolu Saglik Merkezi, Gebze
  - Ege Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
  - Karadeniz Technical University Faculty of Medicine, Trabzon
- United Kingdom (10):
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire
  - Royal United Hospital, Bath
  - University Hospital Birmingham, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Ninewells Hospital - PPDS, Dundee
  - Leicester Royal Infirmary, Leicester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - The Royal Marsden NHS Foundation Trust, Sutton
  - Pinderfields General Hospital, Wakefield

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Puig N, Leleu X, Lee HC, Davies FE, Hajek R, Hungria V, Thompson MA, Cook G, Ojeda JV, Weisel KC, Berdeja JG, Usmani SZ, Symeonidis A, Nascimento-Ferreira I, Arthur D, Mokra L, Ren K, Cherepanov D, Terpos E. Comparative Effectiveness and Safety of PI-Rd Triplets in Relapsed/Refractory Multiple Myeloma: INSIGHT-MM Data Analysis. Eur J Haematol. 2026 Jan 13. doi: 10.1111/ejh.70079. Online ahead of print. PMID 41528195
- [Derived] Rifkin RM, Costello CL, Birhiray RE, Kambhampati S, Richter J, Abonour R, Lee HC, Stokes M, Ren K, Stull DM, Cherepanov D, Bogard K, Noga SJ, Girnius S. In-class transition from bortezomib-based therapy to IRd is an effective approach in newly diagnosed multiple myeloma. Future Oncol. 2024 Jan;20(3):131-143. doi: 10.2217/fon-2023-0272. Epub 2023 Oct 9. PMID 37807952
- [Derived] Thompson MA, Boccadoro M, Leleu X, Vela-Ojeda J, van Rhee F, Weisel KC, Rifkin RM, Usmani SZ, Hajek R, Cook G, Abonour R, Armour M, Morgan KE, Yeh SP, Costello CL, Berdeja JG, Davies FE, Zonder JA, Lee HC, Omel J, Spencer A, Terpos E, Hungria VTM, Puig N, Fu C, Ferrari RH, Ren K, Stull DM, Chari A. Rates of Influenza and Pneumococcal Vaccination and Correlation With Survival in Multiple Myeloma Patients. Clin Lymphoma Myeloma Leuk. 2023 Mar;23(3):e171-e181. doi: 10.1016/j.clml.2022.12.003. Epub 2022 Dec 7. PMID 36641358
- [Derived] Hajek R, Minarik J, Straub J, Pour L, Jungova A, Berdeja JG, Boccadoro M, Brozova L, Spencer A, van Rhee F, Vela-Ojeda J, Thompson MA, Abonour R, Chari A, Cook G, Costello CL, Davies FE, Hungria VT, Lee HC, Leleu X, Puig N, Rifkin RM, Terpos E, Usmani SZ, Weisel KC, Zonder JA, Barinova M, Kuhn M, Silar J, Capkova L, Galvez K, Lu J, Elliott J, Stull DM, Ren K, Maisnar V. Ixazomib-lenalidomide-dexamethasone in routine clinical practice: effectiveness in relapsed/refractory multiple myeloma. Future Oncol. 2021 Jul;17(19):2499-2512. doi: 10.2217/fon-2020-1225. Epub 2021 Mar 26. PMID 33769076
- [Derived] Costello C, Davies FE, Cook G, Vela-Ojeda J, Omel J, Rifkin RM, Berdeja J, Puig N, Usmani SZ, Weisel K, Zonder JA, Terpos E, Spencer A, Leleu X, Boccadoro M, Thompson MA, Romanus D, Stull DM, Hungria V. INSIGHT MM: a large, global, prospective, non-interventional, real-world study of patients with multiple myeloma. Future Oncol. 2019 May;15(13):1411-1428. doi: 10.2217/fon-2019-0013. Epub 2019 Feb 28. PMID 30816809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 130 investigative sites in China, Taiwan, Belgium, France, Germany, Greece, Israel, Italy, Spain, Turkey, United Kingdom, Brazil, Colombia, Mexico, United States from 1 July 2016 to 30 September 2021. A total of 4253 participants were enrolled in this study.
Pre-assignment Details: Prospective data was collected for newly diagnosed multiple myeloma (NDMM) and Relapsed/Refractory multiple myeloma (RRMM) participants. Participants were also divided for analysis of some part of this study according to lines of therapy (LOT) they received. The final outcomes analysis performed at the end of study included 3263 participants excluding 990 participants from 4253 due to concerns around the robustness of data. Participants who received >1 LOT were counted more than once.
Groups:
- Newly Diagnosed (ND) MM: Participants newly diagnosed with MM within 3 months from initiation of treatment were enrolled for 3 years, and followed for at least 2 years, until death, or the end of the study, whichever comes first (up to approximately 5 years).
- Relapsed/Refractory (R/R) MM: Participants diagnosed with RRMM who previously received 1 to 3 prior lines of therapy were enrolled for 3 years, and followed for at least 2 years, until death, or the end of the study, whichever comes first (up to approximately 5 years).
Period: Overall Study
Arm/Group | Newly Diagnosed (ND) MM | Relapsed/Refractory (R/R) MM
Started | 2338 | 1915
1st Line of Therapy (The most common treatment regimens prescribed in participants treated in 1st line of therapy were proteosome inhibitor (PI)+ immunomodulatory drug (IMiD), PI+ alkylating agent (AA), and PI treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years).) | 2193 | 68
2nd Line of Therapy (The most common treatment regimens prescribed in participants treated in 2nd line of therapy were PI+IMiD, IMiD, and PI treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years).) | 928 | 950
3rd Line of Therapy (The most common treatment regimens prescribed in participants treated in 3rd line of therapy were IMiD, PI+IMiD, and monoclonal antibody (mAB)+IMiD treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years).) | 406 | 1049
4th Line of Therapy (The most common treatment regimens prescribed in participants treated in 4th line of therapy were mAb, mAb+IMiD, and mAB+PI treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years).) | 185 | 727
>4th Line of Therapy (The most common treatment regimens prescribed in participants treated in >4th line of therapy were mAb, PI, and IMiD+AA treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years).) | 153 | 767
Line of Therapy: Unknown (Missing line of therapy with respect to recorded regimen or have not observed any regimen with line of therapy on or after study entry. Participants were observed until study discontinuation, death or end of study (up to approximately 5 years).) | 54 | 93
Completed | 0 | 0
Not Completed | 2338 | 1915
Not completed — Too ill to Participate | 13 | 8
Not completed — Patient declined participation and declined follow-up for survival | 34 | 26
Not completed — Patient withdrew consent | 64 | 58
Not completed — Physician discretion | 4 | 8
Not completed — Change in physician or transferred to another treatment center | 72 | 62
Not completed — On Hospice | 20 | 26
Not completed — Deceased | 474 | 642
Not completed — Lost to Follow-up | 73 | 63
Not completed — Due to study discontinued at site | 100 | 85
Not completed — Reason not Specified | 1484 | 937

BASELINE CHARACTERISTICS:
Population: All Enrolled Population included all participants who signed the inform consent form.
Groups:
- NDMM: Participants with newly diagnosed MM within 3 months from initiation of treatment were enrolled for 3 years, and followed for at least 2 years, until death, or the end of the study, whichever comes first (up to approximately 5 years).
- RRMM: Participants diagnosed with RRMM who previously received 1 to 3 prior lines of therapy were enrolled for 3 years, and followed for at least 2 years, until death, or the end of the study, whichever comes first (up to approximately 5 years).
- Total: Total of all reporting groups
Arm/Group | NDMM | RRMM | Total
Number analyzed (Participants) | 2338 | 1915 | 4253
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at study entry was provided by the participant or calculated from date of birth if age was missing as the integer part of: Age (years) = (Informed Consent Date - Date of Birth + 1) / 365.25. Population: Number analyzed are the number of participants available for baseline age continuous.
  years
    number analyzed (Participants) | 2337 | 1914 | 4251
    (all) | 64.7 (10.94) | 66.0 (10.42) | 65.2 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1317 | 1128 | 2445
  Male | 1021 | 787 | 1808
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 348 | 285 | 633
  Not Hispanic or Latino | 1297 | 1004 | 2301
  Unknown or Not Reported | 693 | 626 | 1319
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 230 | 160 | 390
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 153 | 111 | 264
  White | 1506 | 1273 | 2779
  More than one race | 25 | 16 | 41
  Unknown or Not Reported | 424 | 355 | 779

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Co-morbidities
Description: Charlson Comorbidity Index (CCI) was used to represent number of participants with co-morbidities. CCI is a method of categorizing comorbidities of participants. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a participant. A score of 0 = no comorbidities found, 1 = not ill, 2 = mildly ill, 3 = moderately ill, 4 = severely ill, and ≥5 = moribund. The higher the score, the more likely the predicted outcome resulted in mortality or higher resource use.
Time Frame: Baseline up to 5 years
Population: All Enrolled Population included all participants who signed the inform consent form. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- NDMM: Participants newly diagnosed with MM within 3 months from initiation of treatment were enrolled for 3 years, and followed for at least 2 years, until death, or the end of the study, whichever comes first (up to approximately 5 years).
Arm/Group | NDMM | RRMM
Number analyzed (Participants) | 1761 | 1440
Participants
  0-1 | 1279 | 1064
  2-3 | 307 | 247
  4-5 | 66 | 60
  >5 | 38 | 19
  Missing | 71 | 50

2. Primary Outcome: Number of Participants Diagnosed With Newly Diagnosed Multiple Myeloma (NDMM) and Relapsed/Refractory Multiple Myeloma (R/RMM)
Description: Participants diagnosed with NDMM and R/RMM were determined at the start of the study.
Time Frame: At Baseline
Population: All Enrolled Population included all participants who signed the inform consent form.
Measure: Count of Participants; unit: Participants
Arm/Group | NDMM | RRMM
Number analyzed (Participants) | 2338 | 1915
Participants | 2338 | 1915

3. Primary Outcome: Number of Participants Diagnosed With Symptoms of ND MM and R/R MM During the Study
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | NDMM | RRMM
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Sites of Disease Diagnosed With ND MM and R/R MM
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | NDMM | RRMM
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Number of Participants With ECOG (Eastern Cooperative Oncology Group) Performance Status
Description: ECOG-PS measured on-therapy (time between first dose and last dose date with a 30-day lag) assessed participant's performance status on 6 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50% of waking hours), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead. The line of Therapy was determined at study entry.
Time Frame: At Baseline
Population: All Enrolled Population included all participants who signed informed consent. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | NDMM | RRMM
Number analyzed (Participants) | 1761 | 1440
Participants
  Grade 0 | 714 | 710
  Grade 1 | 727 | 559
  Grade 2 | 171 | 113
  Grade 3 | 61 | 22
  Grade 4 | 13 | 2
  Missing | 75 | 34

6. Primary Outcome: Number of Participants With Myeloma Frailty Index
Description: Frailty is defined as the combination of unintentional weight loss, exhaustion, low physical activity, slow walking speed, and muscular weakness. The Myeloma Frailty Index is a composite index that was calculated using the points system, which produces a range of values from 0 to 5. Participants with score 0= fit, score 1= intermediate, and score ≥2= frail. Higher score indicates likeliness that the predicted outcome will result in frailty. The line of Therapy was determined at study entry.
Time Frame: At Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- 1st Line of Therapy: The most common treatment regimens prescribed in participants treated in 1st line of therapy were PI+IMiD, PI+AA, and PI treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years).
- 2nd Line of Therapy: The most common treatment regimens prescribed in participants treated in 2nd line of therapy were PI+IMiD, IMiD, and PI treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years).
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy
Number analyzed (Participants) | 1761 | 1440
Participants
  0: Fit | 517 | 428
  1: Intermediate | 218 | 202
  ≥2: Frail | 190 | 130
  Missing | 836 | 680

7. Primary Outcome: Number of Participants Evaluated for Minimal Residual Disease (MRD)
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | NDMM | RRMM
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Number of Participants Evaluated for Gene Expression Profiling (GEP)
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | NDMM | RRMM
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Number of Participants Evaluated for Cytogenetics Using Fluorescence in Situ Hybridization (FISH)
Description: FISH methodology was reported with Yes/No results for the following tests: deletion (17p)/p53 [Del(17p)/p53], translocation (4,14) [t(4,14)], and translocation (14,16) [t(14,16)].
Time Frame: At Baseline
Population: All Enrolled Population included all participants who signed the inform consent form, out of which 990 participants were excluded during the final analysis due to concerns around robustness of data. The data is reported as per the known line of therapies. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- 3rd Line of Therapy: The most common treatment regimens prescribed in participants treated in 3rd line of therapy were IMiD, PI+IMiD, and mAB+IMiD treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years).
- 4th Line of Therapy: The most common treatment regimens prescribed in participants treated in 4th line of therapy were mAb, mAb+IMiD, and mAB+PI treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years).
- >4th Line of Therapy: The most common treatment regimens prescribed in participants treated in >4th line of therapy were mAb, PI, and IMiD+AA treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years).
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 1790 | 686 | 458 | 249 | 80
Participants
  Del(17p)/p53: Not Reported/Performed | 208 | 20 | 7 | 4 | 0
  Del(17p)/p53: Yes | 126 | 23 | 12 | 5 | 0
  Del(17p)/p53: No | 950 | 147 | 55 | 24 | 12
  Del(17p)/p53: Not Done - Inferred | 399 | 17 | 2 | 2 | 0
  Del(17p)/p53: Missing | 107 | 479 | 382 | 214 | 68
  t(4,14): Not Reported/Performed | 208 | 20 | 7 | 4 | 0
  t(4,14): Yes | 116 | 24 | 4 | 5 | 3
  t(4,14): No | 957 | 144 | 63 | 25 | 9
  t(4,14): Not Done - Inferred | 401 | 18 | 2 | 2 | 0
  t(4,14): Missing | 108 | 480 | 382 | 213 | 68
  t(14,16): Not Reported/Performed | 208 | 20 | 7 | 4 | 0
  t(14,16): Yes | 50 | 7 | 0 | 3 | 0
  t(14,16): No | 1007 | 157 | 67 | 27 | 12
  t(14,16): Not Done - Inferred | 416 | 18 | 2 | 2 | 0
  t(14,16): Missing | 109 | 484 | 382 | 213 | 68

10. Primary Outcome: Number of Participants Evaluated for International Staging System (ISS)/ Revised (R)-ISS Stage
Description: ISS disease stages were defined as I:low risk, β2-Microglobulin<3.5mg/L, albumin≥3.5g/dL, II:not stage I or III, III:high risk,β2-Microglobulin≥5.5mg/L). R-ISS is based on ISS, chromosomal abnormalities (CA), and lactate dehydrogenase (LDH). R-ISS disease stages were defined as I: ISS Stage I and standard risk CA by FISH and normal LDH (i.e. <=300 U/L), II: Neither R-ISS Stage I nor Stage III, III: ISS Stage III and either high risk CA by FISH or high LDH (i.e. >300 U/L).
Time Frame: At Baseline
Population: All Enrolled Population included all participants who signed informed consent. Overall number of participants are the number of participants available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | NDMM | RRMM
Number analyzed (Participants) | 1761 | 1440
Participants
  ISS Stage I | 395 | 236
  ISS Stage II | 387 | 267
  ISS Stage III | 520 | 297
  ISS Not Available | 138 | 376
  ISS Missing | 321 | 264
  R-ISS Stage I | 127 | 40
  R-ISS Stage II | 319 | 145
  R-ISS Stage III | 76 | 24
  R-ISS Not available | 69 | 285
  R-ISS Missing | 1170 | 946

11. Primary Outcome: Duration of Treatment for Participants With and Without Stem Cell Transplant
Description: Data was analyzed for participants with and without stem cell transplant for all enrolled population, included all participants who signed the inform consent form, out of which 990 participants were excluded during the final analysis due to concerns around robustness of data.
Time Frame: Baseline up to 5 years
Population: All Enrolled Population included all participants who signed the inform consent form, out of which 990 participants were excluded during the final analysis due to concerns around robustness of data. Overall number analyzed are the number of participants with data available for analyses. The data is reported as per the known line of therapies.
Measure: Median (Full Range); unit: months
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 1597 | 575 | 390 | 227 | 77
months | 4.5 [0 to 45] | 6.4 [0 to 57] | 9.2 [0 to 80] | 11.5 [0 to 68] | 11.5 [0 to 52]

12. Primary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the number of months from the index regimen start date within each line of therapy, starting with the line during study entry, until the date of death. The Kaplan Meier estimates was used for the analysis.
Time Frame: Baseline up to 5 years
Population: All Enrolled Population, included all participants who signed the inform consent form, out of which 990 participants were excluded during the final analysis due to concerns around robustness of data. The data is reported as per the known line of therapies. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 1790 | 1331 | 1050 | 739 | 453
months | NA [NA to NA] — Median and 95% confidence interval (CI) was not estimable due to an insufficient number of participants with events of death. | 47.67 [45.34 to NA] — The upper limit of CI was not estimable due to an insufficient number of participants with events of death. | 32.07 [26.84 to 39.56] | 20.60 [17.51 to 23.36] | 13.44 [10.91 to 15.90]

13. Primary Outcome: Disease Progression Status on Each Regimen
Description: Disease progression status was assessed by physician interpretation of IMWG Response criteria.
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Groups:
- Unknown: Missing line of therapy with respect to recorded regimen or have not observed any regimen with line of therapy on or after study entry. Participants were observed until study discontinuation, death or end of study (up to approximately 5 years).
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy | Unknown
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Response to Each Regimen
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy | Unknown
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Time to Next Therapy
Description: The line of Therapy was determined at study entry. The Kaplan Meier estimates was used for the analysis.
Time Frame: Baseline up to 5 years
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 1790 | 1331 | 1050 | 739 | 453
months | 30.39 [26.87 to 33.74] | 15.44 [13.63 to 17.08] | 9.46 [8.34 to 10.81] | 6.90 [6.11 to 7.82] | 5.95 [5.16 to 6.70]

16. Primary Outcome: Number of Participants With Stem Cell Transplant
Time Frame: Baseline up to 5 years
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 1790 | 686 | 458 | 249 | 80
Participants | 1790 | 686 | 458 | 249 | 80

17. Secondary Outcome: Number of Participants Receiving Different Treatment Combinations
Time Frame: Baseline up to 5 years
Population: All Enrolled Population included all participants who signed the inform consent form. Participants were reported more than once in each line of therapy. Data is reported only for 1st, 2nd 3rd and 4th line of therapy. The overall number of participants analyzed is the number of participants available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy
Number analyzed (Participants) | 2195 | 1685 | 1279 | 845
Participants
  Bortezomib and Lenalidomide (VR) | 560 | 86 | 19 | 10
  Bortezomib and Cyclophosphamide (VC) | 497 | 99 | 43 | 18
  Bortezomib and Thalidomide (VT) | 272 | 60 | 10 | 11
  Bortezomib and Melphalan (VM) | 75 | 16 | 8 | 3
  Lenalidomide (R) | 21 | 39 | 22 | 5
  Lenalidomide and Dexamethasone (RD) | 86 | 218 | 126 | 30
  Cyclophosphamide and Thalidomide (CT) | 60 | 37 | 11 | 5
  Melphalan and Thalidomide (MT) | 10 | 3 | 4 | 3
  Thalidomide and Dexamethasone (TD) | 7 | 1 | 5 | 2
  Bortezomib and dexamethasone (VD) | 95 | 47 | 18 | 6
  Ixazomib and Lenalidomide (IR) | 4 | 96 | 115 | 34
  Carfilzomib and Lenalidomide (KR) | 63 | 112 | 42 | 18
  Bortezomib and Pomalidomide (VPom) | 0 | 7 | 2 | 6
  Carfilzomib and Pomalidomide (KPom) | 1 | 27 | 22 | 12
  Carfilzomib and dexamethasone (KD) | 3 | 59 | 76 | 46
  Daratumumab-Bortezomib (dara-V) | 7 | 110 | 78 | 46
  Daratumumab-Ixazomib (dara-I) | 1 | 12 | 7 | 3
  Daratumumab-Lenalidomide (dara-R) | 3 | 149 | 70 | 31
  Daratumumab-Pomalidomide (dara-Pom) | 0 | 49 | 72 | 43
  Ixazomib and Dexamethasone (ID) | 1 | 14 | 13 | 9
  Ixazomib (I) | 0 | 6 | 5 | 4
  Pomalidomide and Dexamethasone (PomD) | 0 | 12 | 66 | 39
  Daratumumab (Dara) | 0 | 15 | 21 | 56
  Elotuzumab and Lenalidomide (Elo-R) | 7 | 42 | 20 | 10
  Elotuzumab-Pomalidomide (Elo-Pom) | 0 | 6 | 10 | 14
  Elotuzumab-Other Regimen (Elo-Other) | 6 | 4 | 4 | 1
  Other Regimen | 416 | 359 | 390 | 380

18. Secondary Outcome: Number of Treatment Sequencing
Description: Drug classes were based on the earliest regimen in each corresponding Line of Therapy. The data for this outcome measure was analyzed as per line of therapy.
Time Frame: Baseline up to 5 years
Population: All Enrolled Population included all participants who signed informed consent. Participants were reported more than once in each line of therapy. Data is reported only for 1st, 2nd and 3rd line of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy
Number analyzed (Participants) | 4224 | 2748 | 1734
Participants
  mAB based | 41 | 77 | 129
  mAB/IMID based | 290 | 213 | 128
  mAB/PI based | 156 | 119 | 69
  mAB/alkalytor based | 2 | 7 | 6
  mAB/IMID/PI based | 36 | 14 | 12
  Cytotoxic | 74 | 59 | 49
  IMID based | 515 | 361 | 118
  PI based | 366 | 204 | 101
  Alkylator based | 79 | 40 | 33
  PI/IMID based | 608 | 295 | 115
  PI/alkylator based | 351 | 137 | 57
  IMID/alkylator based | 123 | 119 | 57
  PI/IMID/alkylator based | 34 | 14 | 7
  Other | 59 | 32 | 46
  Unknown | 1490 | 1057 | 807

19. Secondary Outcome: Number of Participants in the Treatment Rechallenge
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Clinical Outcomes for Different Strategies
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Clinical Outcomes Between Continuous Treatment and Intermittent Treatment Strategy
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Triggers of Treatment Initiation at Relapse Including Biochemical Progression or Symptomatic Progression
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Reasons for Treatment Modifications
Time Frame: Baseline up to 5 years
Population: All Enrolled Population included all participants who signed informed consent. Participants received more than one LOT and are counted in more than one LOT. The data is reported as per the known line of therapies. Participants were counted multiple times in different categories. The overall number of participants analyzed is the number of participants available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 2260 | 1878 | 1416 | 700 | 500
Participants
  Adverse Event Related to Drug | 920 | 676 | 459 | 240 | 187
  Other | 425 | 333 | 248 | 110 | 81
  Planned Change | 386 | 274 | 205 | 99 | 62
  Adverse Event Not Related to MM Therapy Drug | 234 | 243 | 179 | 91 | 62
  Current Dose Tolerated, Dose Increased | 110 | 107 | 105 | 47 | 30
  Dose Delay Due to Toxicity | 63 | 91 | 65 | 32 | 22
  Patient/Family Preference | 53 | 58 | 39 | 19 | 16
  Treatment Fatigue | 25 | 36 | 33 | 17 | 13
  Lack of Response | 16 | 23 | 27 | 11 | 13
  COVID-19 Restrictions | 13 | 21 | 22 | 11 | 8
  Relapse - Biochemical Progression | 9 | 17 | 19 | 11 | 7
  COVID-19 Diagnosis (Confirmed Positive) | 5 | 11 | 7 | 8 | 3
  Relapse - Symptomatic/Clinical Progression | 5 | 10 | 3 | 2 | 3
  COVID-19 Diagnosis (Suspected Positive) | 3 | 0 | 1 | 0 | 0
  Missing | 6 | 13 | 4 | 2 | 1

24. Primary Outcome: Number of Participants With Global Health Status Scale/Quality of Life (QoL) Among MM Participants
Description: The Global Health Status scale/QoL scale included 2 questions measured with a 7-point numeric rating scale (very poor to excellent). Raw scores are converted into scale scores ranging from 0 to 100. A higher score represents better HRQoL.
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy | Unknown
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Healthcare Resource Utilization (HRU) Among MM Participants
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Associations Between Presentation and Disease Characteristics
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Associations Between Choice Of Therapy and Clinical Outcomes
Time Frame: Baseline up to 5 years
Population: As the study was early terminated data was not collected for this outcome measure.
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Number of Participants With Atleast One Treatment-emergent Adverse Events Leading to Treatment Discontinuation
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. Treatment discontinuation includes temporary and permanent discontinuation, drug modification, and second primary malignancies.
Time Frame: Baseline up to 5 years
Population: Participants who received Takeda products and signed informed consent form were included in the analysis. As pre-specified in SAP, data for treatment-emergent adverse events was planned to be collected and reported for Takeda products only. Participants were counted more than once in each line of therapy towards the total. The data is reported as per the known line of therapies.
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy
Number analyzed (Participants) | 2261 | 1878 | 1455 | 912 | 500
Participants | 375 | 275 | 178 | 98 | 95

ADVERSE EVENTS:
Time Frame: From start of study, until death, or the end of the study, whichever comes first (up to 5 years)
Description: As per planned analysis,mortality was collected for all participants; serious/other adverse events were collected only for participants who signed an informed consent form and had robust data. Data was reported per line of therapies and robustness concerns.As pre-specified in SAP,serious and other adverse events were collected and reported for Takeda products only.A participant maybe counted across multiple lines of therapy, allowing same participant to be represented in multiple index regimens.
Groups:
- Robustness Concerns: 1st Line of Therapy: The most common treatment regimens prescribed in participants treated in 1st line of therapy were PI+IMiD, PI+AA, and PI treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years). Only participants treated in 1st line of therapy with concerns around the robustness of data were included in this arm.
- Robustness Concerns: 2nd Line of Therapy: The most common treatment regimens prescribed in participants treated in 2nd line of therapy were PI+IMiD, IMiD, and PI treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years). Only participants treated in 2nd line of therapy with concerns around the robustness of data were included in this arm.
- Robustness Concerns: 3rd Line of Therapy: The most common treatment regimens prescribed in participants treated in 3rd line of therapy were IMiD, PI+IMiD, and mAB+IMiD treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years). Only participants treated in 3rd line of therapy with concerns around the robustness of data were included in this arm.
- Robustness Concerns: 4th Line of Therapy: The most common treatment regimens prescribed in participants treated in 4th line of therapy were mAb, mAb+IMiD, and mAB+PI treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years). Only participants treated in 4th line of therapy with concerns around the robustness of data were included in this arm.
- Robustness Concerns: >4th Line of Therapy: The most common treatment regimens prescribed in participants treated in >4th line of therapy were mAb, PI, and IMiD+AA treatment as part of their index regimen while enrolled in the study and were observed until study discontinuation, death or end of study (up to approximately 5 years). Only participants treated in >4th line of therapy with concerns around the robustness of data were included in this arm.
- Robustness Concerns: Unknown Line of Therapy: The 'Unknown Line of Therapy' indicates either: 1) participant was on a regimen on or after study entry, but missing line of therapy with respect to that regimen or 2) have not observed any regimen with line of therapy on or after study entry. Only participants in unknown line of therapy with concerns around the robustness of data were included in this arm.
Arm/Group | 1st Line of Therapy | 2nd Line of Therapy | 3rd Line of Therapy | 4th Line of Therapy | >4th Line of Therapy | Robustness Concerns: 1st Line of Therapy | Robustness Concerns: 2nd Line of Therapy | Robustness Concerns: 3rd Line of Therapy | Robustness Concerns: 4th Line of Therapy | Robustness Concerns: >4th Line of Therapy | Robustness Concerns: Unknown Line of Therapy
All-Cause Mortality (participants affected / at risk) | 351/1790 | 418/1331 | 420/1050 | 348/739 | 234/453 | 58/340 | 72/303 | 65/222 | 32/86 | 6/24 | 28/147
Serious Adverse Events (participants affected / at risk) | 269/1849 | 101/773 | 82/455 | 43/239 | 38/181 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 306/1849 | 125/773 | 79/455 | 39/239 | 32/181 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 1st Line of Therapy (N=1849) | 2nd Line of Therapy (N=773) | 3rd Line of Therapy (N=455) | 4th Line of Therapy (N=239) | >4th Line of Therapy (N=181) | Robustness Concerns: 1st Line of Therapy (N=0) | Robustness Concerns: 2nd Line of Therapy (N=0) | Robustness Concerns: 3rd Line of Therapy (N=0) | Robustness Concerns: 4th Line of Therapy (N=0) | Robustness Concerns: >4th Line of Therapy (N=0) | Robustness Concerns: Unknown Line of Therapy (N=0)
Anaemia (Blood and lymphatic system disorders) | 6 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 5 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 1 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 9 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Microvascular coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parathyroid disorder (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic duct obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 10 | 3 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder volvulus (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 5 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 42 | 17 | 17 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 3 | 5 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 8 | 4 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis syndrome (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 6 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteochondral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Human metapneumovirus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza A virus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respirovirus test positive (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotavirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rubulavirus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autonomic neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post stroke seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device loosening (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 10 | 3 | 4 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toe amputation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0/0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1st Line of Therapy (N=1849) | 2nd Line of Therapy (N=773) | 3rd Line of Therapy (N=455) | 4th Line of Therapy (N=239) | >4th Line of Therapy (N=181) | Robustness Concerns: 1st Line of Therapy (N=0) | Robustness Concerns: 2nd Line of Therapy (N=0) | Robustness Concerns: 3rd Line of Therapy (N=0) | Robustness Concerns: 4th Line of Therapy (N=0) | Robustness Concerns: >4th Line of Therapy (N=0) | Robustness Concerns: Unknown Line of Therapy (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 5 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 16 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 14 | 14 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Systolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dacryoadenitis acquired (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aerophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal dilatation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 13 | 7 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 14 | 13 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 7 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 25 | 10 | 8 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperpyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 11 | 4 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 8 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunosuppression (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral allergy syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 5 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Candida sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 6 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pustule (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 5 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenovirus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis E virus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 4 | 3 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autonomic neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 8 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Formication (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 64 | 31 | 15 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 43 | 9 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 6 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile erythema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 10 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculovesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 3 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was terminated 3 years early due to business reprioritization within Takeda.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT02761187/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT02761187/SAP_001.pdf